CLINICAL TRIAL: NCT03043222
Title: Effect of Prostatic Urethral Lift (PUL) Versus Prostate Arterial Embolization (PAE),Novel Minimally Invasive Treatment Options on Health-related Quality of Life (HRQoL) in Men With Lower Urinary Tract Symptoms Secondary to BPH.
Brief Title: Innovative Minimally Invasive Options in Treatment of Urinary Problems Related to Prostate Enlargement (BPH) in Men
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn from IRB
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Keith Pereira, MD:, MD, Assistant professor, Interventional Radiology, St. Louis University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27936
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia; Urinary Frequency/Urgency; Urinary Incontinence, Urge; Incontinence, Urinary; Nocturia
Keywords: prostate artery embolization; Prostatic Urethral Lift, Urolift; Minimally invasive; non-surgical; maintenance of sexual function; complications of TURP , surgery
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia; Urinary Incontinence, Urge; Urinary Incontinence; Nocturia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- PAE-Prostate Arterial Embolization (Experimental): PAE-Prostate Arterial Embolization
  Interventions: Device: UroLift as artifical device for prostatic urethral lift.; Device: Embospheres Microspheres as embolic agents for prostate artery embolization
- PUL- Prostatic urethral lift (Active Comparator): PUL- Prostatic urethral lift
  Interventions: Device: UroLift as artifical device for prostatic urethral lift.; Device: Embospheres Microspheres as embolic agents for prostate artery embolization

INTERVENTIONS:
Device: UroLift as artifical device for prostatic urethral lift. — UroLift as artifical device for prostatic urethral lift. The PUL treatment is a minimally invasive approach to treating an enlarged prostate, or BPH, that lifts or holds the enlarged prostate tissue using clips so that it is out of the way so it no longer blocks the urethra. There is no cutting, heating or removal of prostate tissue.
  Other Names: Prostatic urethral lift.
Device: Embospheres Microspheres as embolic agents for prostate artery embolization — Embospheres Microspheres as embolic agents for prostate artery embolization Arterial access will be obtained.Under live X-ray monitoring and using contrast, a catheter will be advanced into the artery to the prostate gland.Small micro spherical particles (Embopheres Microspheres) will be injected though the catheter to occlude the artery and cut off blood supply to the enlarged prostate. The prostate is then expected to shrink , thus relieving urinary symptoms related to prostate enlargement.There is no cutting or removal of prostate tissue.Once the procedure is complete, in case of wrist access compression will be achieved with a band; in case of groin access a closure device will be used to plug the site of entry.
  Other Names: Prostate artery embolization

SUMMARY:
For ageing men, Health related quality of life ( HRQoL) is challenged by two common issues: the onset of bothersome urinary symptoms attributable to prostate enlargement and diminishing ability to maintain normal sexual activity and function; both issues are important to men, yet often the treatment of the former has adverse effects on the latter. Current medical and surgical treatments offer symptomatic improvement of urinary symptoms. However long recovery times, degradation of sexual function and incontinence may negatively affect a patient's QoL.

Prostatic urethral lift (PUL) and prostate artery embolization (PAE) represent two evolving techniques with contrasting mechanisms of action (mechanical decompression vs angiographic embolization). Both are minimally invasive, yield relief of urinary symptoms and have similar safety profiles. More importantly neither causes degradation of sexual function or urinary continence. Although multiple studies are being reported on PUL and PAE alike, currently there are no prospective clinical trials comparing these two technologies. We aim to prospectively evaluate and compare HRQol outcomes of PUL and PAE. Results of this study could have a great impact on patient outcomes in men opting for minimally invasive, sexual function sparing treatment options for symptom relief from prostate enlargement.

DETAILED DESCRIPTION:
As the population ages, there is a growing need to find ways for people to live longer with satisfactory quality of life (QoL), even in the midst of increasing health problems. For the ageing man, Health related quality of life ( HRQoL) is challenged by two common issues: the onset of bothersome LUTS attributable to benign prostatic hypertrophy (BPH) and diminishing ability to maintain normal sexual activity and function; both issues are important to men, yet often the treatment of the former has adverse effects on the latter.

Current medical and surgical treatments like TURP for BPH offer symptomatic improvement of LUTS but may adversely affect a patient's QOL and satisfaction. Peri-operative complications and long recovery times, degradation of sexual function and iatrogenic incontinence may negatively affect a patient's QoL overall, resulting in patient viewing this as a treatment failure. Therefore when evaluating treatment options for BPH, treatment options with important QOL measures of satisfaction have to be considered.

Prostatic urethral lift (PUL) and prostate artery embolization (PAE) represent two evolving techniques with contrasting mechanisms of action (mechanical decompression vs angiographic embolization). Multiple prospective and retrospective studies have shown that both PUL and PAE yield relief of lower urinary tract symptoms over a period of several weeks. They display similar safety profiles with self-limiting pelvic discomfort characterizing the commonest minor adverse event. Both procedures are minimally invasive and have the potential to be carried out under local anesthesia and in the outpatient setting with suitability for patients with cardiovascular comorbidities. Another important finding is that neither has been found to cause degradation of sexual function.

Although there are an increasing number of data series being reported on PUL and PAE alike, currently there are no prospective clinical trials comparing these two technologies. We aim to prospectively evaluate and compare HRQol outcomes of PUL and PAE. All the endpoints will be evaluated using validated questionnaires and laboratory values. Results of this study will be transferable to clinical practice and could have a great impact on patient outcomes in men opting for minimally invasive, sexual function sparing treatment options for symptom relief from LUTS due to BPH in all practice settings.

ELIGIBILITY:
Inclusion Criteria:

Male aged ≥40 yr Willing, able and mentally competent to provide written informed consent and willing to comply with all study procedures and be available for the duration of the study Diagnosis of urinary symptoms (LUTS) from prostatic enlargement (BPH) refractory to medical therapy for at least 6 months.

International Prostate Symptom Score >12

Exclusion Criteria:

* PUL

  1. Active urinary tract infections, prostatitis, or interstitial cystitis.
  2. Biopsy proven prostate, bladder, or urethral cancer.

     The following patients must undergo prostate biopsy with a minimum of 12 cores and have a negative histopathology report to be enrolled in the study:
     * Patients with digital rectal examination (DRE) findings suspicious for prostate cancer
     * Patients with baseline PSA levels > 10 ng/mL
     * Patients with baseline PSA levels >2.5 ng/mL and < 10ng/mL AND free PSA < 25% of total PSA Patients with cystoscopy findings suspicious for bladder cancer must undergo biopsy and have a negative histopathology report to be enrolled in the study
  3. Significant median lobe enlargement.
  4. Large prostates, volume >80 g.
  5. Bladder atonia, neurogenic bladder disorder or other neurological disorder that is impacting bladder function (e.g. multiple sclerosis, Parkinson's disease, spinal cord injuries, etc.)
  6. Urethral stricture, bladder neck contracture, sphincter abnormalities, bladder diverticulum, urinary obstruction due to causes other than BPH, or other potentially confounding bladder or urethral disease or condition
  7. Urethral conditions that may prevent insertion of a rigid 20F cystoscope
  8. Current urinary retention.
  9. Acontractile detrusor.
  10. Current gross hematuria
  11. Known upper tract renal disease
  12. Cystolithiasis
  13. ASA > 3 or severe medical debilitating condition
  14. History of pelvic irradiation or radical pelvic surgery
  15. Known allergy to nickel.

      PAE
  16. Active urinary tract infections, prostatitis, or interstitial cystitis.
  17. Biopsy proven prostate, bladder, or urethral cancer.

      The following patients must undergo prostate biopsy with a minimum of 12 cores and have a negative histopathology report to be enrolled in the study:
      * Patients with digital rectal examination (DRE) findings suspicious for prostate cancer
      * Patients with baseline PSA levels > 10 ng/mL
      * Patients with baseline PSA levels >2.5 ng/mL and < 10ng/mL AND free PSA < 25% of total PSA Patients with cystoscopy findings suspicious for bladder cancer must undergo biopsy and have a negative histopathology report to be enrolled in the study
  18. Unable to have CT angio of the prostate imaging
  19. Bladder atonia, neurogenic bladder disorder or other neurological disorder that is impacting bladder function (e.g. multiple sclerosis, Parkinson's disease, spinal cord injuries, etc.)
  20. Urethral stricture, bladder neck contracture, sphincter abnormalities, bladder diverticulum, urinary obstruction due to causes other than BPH, or other potentially confounding bladder or urethral disease or condition
  21. Acontractile detrusor.
  22. Known upper tract renal disease
  23. Cystolithiasis
  24. Any known condition that limits catheter-based intervention or is a contraindication to embolization, such as intolerance to a vessel occlusion procedure or severe atherosclerosis. Known major iliac arterial occlusive disease
  25. ASA > 3 or severe medical debilitating condition
  26. Baseline serum creatinine level > 1.8 mg/dl
  27. Previous rectal surgery other than hemorrhoidectomy, or history of rectal disease
  28. History of pelvic irradiation or radical pelvic surgery
  29. Allergy to iodinated contrast agents

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in QOL | 3,6,12 months
  Improvement in QOL score

SECONDARY OUTCOMES:
Number of patients with clinical adverse events | 1 day, 8 days and 1,3,6,12 months
  Short and medium term complications assessed by Clavien-Dindo Classification of Surgical Complications
Post operative morbidity | 1 day, 8 days and 1 month
  Morbidity (Intraprocedural and periprocedural data): Pain, hematuria, Procedure time, radiation parameters, duration of post procedure catheterization and hospitalization
Recovery experience | 1 day, 8 days and 1 month
  Recovery experience based on Quality of life (QoL) Visual Analog Scale( VAS)
Improvement in symptoms of LUTS | 3,6,12 months
  Reduction in International Prostate Symptom Score (IPSS) compared to baseline
Lack of change in sexual function | 3,6,12 months
  Reduction of Sexual Health Inventory For Men (SHIM) score compared to baseline
Lack of change in ejaculation during sex | 3,6,12 months
  Change in Male Sexual Health Questionnaire to assess ejaculatory dysfunction (MSHQ-EjD)
Lack of change in urinary incontinence | 3,6,12 months
  Change in Incontinence severity index (ISI) score
Change in Urinary flow after procedure | 3,6,12 months
  Change in Urinary maximal flow rate (Qmax) measured in ml/s on uroflowmetry.
Change in Prostate volume after procedure | 3,6,12 months
  Change in Prostate volume measured in cm3
Change in residual urine left in bladder after procedure | 3,6,12 months
  Change in Postvoid residual urine volume measured in ml
Change in Prostatic specific antigen (PSA) after procedure | 3,6,12 months
  Change in PSA level measured in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Keith Pereira, MD, Principal Investigator — Saint Louis University Hospital; Beneranda Sophia Ford-Glanton, MD, Principal Investigator — Saint Louis University Hospital
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McVary KT, Roehrborn CG, Avins AL, Barry MJ, Bruskewitz RC, Donnell RF, Foster HE Jr, Gonzalez CM, Kaplan SA, Penson DF, Ulchaker JC, Wei JT. Update on AUA guideline on the management of benign prostatic hyperplasia. J Urol. 2011 May;185(5):1793-803. doi: 10.1016/j.juro.2011.01.074. Epub 2011 Mar 21. PMID 21420124
- [Result] Roehrborn CG, Rukstalis DB, Barkin J, Gange SN, Shore ND, Giddens JL, Bolton DM, Cowan BE, Cantwell AL, McVary KT, Te AE, Gholami SS, Moseley WG, Chin PT, Dowling WT, Freedman SJ, Incze PF, Coffield KS, Borges FD, Rashid P. Three year results of the prostatic urethral L.I.F.T. study. Can J Urol. 2015 Jun;22(3):7772-82. PMID 26068624
- [Result] Sonksen J, Barber NJ, Speakman MJ, Berges R, Wetterauer U, Greene D, Sievert KD, Chapple CR, Montorsi F, Patterson JM, Fahrenkrug L, Schoenthaler M, Gratzke C. Prospective, randomized, multinational study of prostatic urethral lift versus transurethral resection of the prostate: 12-month results from the BPH6 study. Eur Urol. 2015 Oct;68(4):643-52. doi: 10.1016/j.eururo.2015.04.024. Epub 2015 Apr 30. PMID 25937539
- [Result] Pisco JM, Rio Tinto H, Campos Pinheiro L, Bilhim T, Duarte M, Fernandes L, Pereira J, Oliveira AG. Embolisation of prostatic arteries as treatment of moderate to severe lower urinary symptoms (LUTS) secondary to benign hyperplasia: results of short- and mid-term follow-up. Eur Radiol. 2013 Sep;23(9):2561-72. doi: 10.1007/s00330-012-2714-9. Epub 2013 Jan 31. PMID 23370938
- [Result] Bagla S, Martin CP, van Breda A, Sheridan MJ, Sterling KM, Papadouris D, Rholl KS, Smirniotopoulos JB, van Breda A. Early results from a United States trial of prostatic artery embolization in the treatment of benign prostatic hyperplasia. J Vasc Interv Radiol. 2014 Jan;25(1):47-52. doi: 10.1016/j.jvir.2013.09.010. Epub 2013 Oct 28. PMID 24176946
- [Result] Uflacker AB, Haskal ZJ. Internal Iliac Artery Embolization for Benign Prostatic Hyperplasia? First Read the Fine Print. J Vasc Interv Radiol. 2015 Sep;26(9):1311-2. doi: 10.1016/j.jvir.2015.06.024. No abstract available. PMID 26314640
- [Result] Pisco JM, Bilhim T, Pinheiro LC, Fernandes L, Pereira J, Costa NV, Duarte M, Oliveira AG. Medium- and Long-Term Outcome of Prostate Artery Embolization for Patients with Benign Prostatic Hyperplasia: Results in 630 Patients. J Vasc Interv Radiol. 2016 Aug;27(8):1115-22. doi: 10.1016/j.jvir.2016.04.001. Epub 2016 Jun 16. PMID 27321890